CLINICAL TRIAL: NCT01110512
Title: Comparative Efficacy of Two Preparations of the Association Diosmin (450 mg) + Hesperidin (50 mg) in the Treatment of Chronic Venous Insufficiency (CVI)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azidus Brasil (Industry)
Responsible Party: Alexandre Frederico, LAL Clinica Pesquisa e Desenvolvimento Ltda
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FLANEO0210; Version 3
Record Dates: First submitted 2010-04-19; First posted 2010-04-26 (Estimated); Last update posted 2010-10-27 (Estimated); Status verified 2010-04

CONDITIONS: Venous Insufficiency
Keywords: Improvement of CVI parameters
MeSH Terms: conditions — Venous Insufficiency | interventions — Diosmin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Flavonid (Experimental)
  Interventions: Drug: Flavonid
- Daflon (Active Comparator)
  Interventions: Drug: Daflon

INTERVENTIONS:
Drug: Flavonid — Diosmin (450 mg) + hesperidin (50 mg)
  1 tablet, 2 times per day.
  Arms: Flavonid
Drug: Daflon — Diosmin (450 mg) + hesperidin (50 mg)
  1 tablet, 2 times per day
  Arms: Daflon

SUMMARY:
It is hoped that with the use of medication, occurs improvement of the CVI parameters, such as edema, pain, night cramps, functional discomfort, heavy feeling and that the drug test is non-inferior than the comparator.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who agree to the terms described in IC;
* Subjects of both genders, aged ≥ 18 and ≤ 75 years with IVC framework of the lower limbs;
* Subjects with CVI ranked 3 to 5, according to CEAP scale;
* Patients complaining of pain and swelling in the lower limbs secondary to IVC;
* Subjects with good mental health that can respond adequately to the study questionnaires;
* Subjects who agree to make any return visits for evaluation;

Exclusion Criteria:

* Patients with CVI classified as 0, 1, 2 or 6, according to CEAP;
* Subjects who have received treatment for varicose veins as laser, medication use topical or oral (eg: brown India, coumarin, and etc.). And surgery in the 03 months preceding the study;
* Patients with other diseases that may interfere with the study results: thrombosis, coagulation disorders and other diseases that the medical criteria, are important to be excluded;
* Pregnant or nursing women;
* Presence of any medical condition that, according to the investigator, should prevent the patient from the study;
* Participation in clinical trials in the twelve months preceding the study;
* Patients with serious illnesses and uncontrolled that need multidrug treatment;
* Patients on diuretics of any kind, regardless of pathology (hypertension, renal or liver disease);
* Values of laboratory tests appropriate security; the Hemoglobin <10 mg / mL the creatinine> 1.5 mg / mL; AST, ALT, GGT ≥ 2 times normal values; the platelet count below 90.000/ml; Total Bilirubin and the fractions ≤ 1.5 times the normal range.
* past medical history of hypersensitivity to drugs of the same pharmacological classes of substances under investigation;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-12 (Estimated); Study Completion 2011-03 (Estimated)

PRIMARY OUTCOMES:
Improvement of the parameters of CVI, such as edema of lower members. | 90 days.
  There will be 06 planned visits (V0, V1, V2, V3, V4 and V5).

SECONDARY OUTCOMES:
Improvement of the parameters of CVI. | 90 days
  There will be 06 planned visits (V0, V1, V2, V3, V4 and V5). Assessment of improvement of signs and symptoms secondary to IVC, which are:
  * paresthesia (tingling);
  * Itching;
  * Pain;
  * cramps at night;
  * Discomfort functional;
  * Heaviness.

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Frederico, Doctor, Principal Investigator — LAL Clinical Reseach e Development Ltda
Locations (1):
- Lal Clínica Pesquisa e Desenvolvimento Ltda, Valinhos, São Paulo, Brazil